CLINICAL TRIAL: NCT00196781
Title: Treatment Decision Making in Early-Stage Prostate Cancer: Evaluation of Computer Based Patient Education and an Interactive Decision Aid
Brief Title: Treatment Decision Making in Early-Stage Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Kathryn L. Taylor, PhD, Principal Investigator, Georgetown University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAMD17-02-1-0062
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Localized Prostate Cancer
Keywords: prostate cancer treatment; medical decision making; informed decision making; shared decision making; decision aid; patient education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the Information + Decision Aid group (Experimental)
  Interventions: Behavioral: CD-ROM-based prostate ca treatment education+decision tools
- Information Only group (Active Comparator)
  Interventions: Behavioral: CD-ROM-based prostate cancer treatment education

INTERVENTIONS:
Behavioral: CD-ROM-based prostate cancer treatment education — The goal was to explore men's use of a CD-ROM-based decision aid for early-stage PCa treatment decisions.
  Other Names: Prostate Cancer Treatment Education
  Arms: Information Only group
Behavioral: CD-ROM-based prostate ca treatment education+decision tools — The goal of the present study was to explore men's use of a CD-ROM-based decision aid for early-stage PCa treatment decisions.
  Other Names: Prostate Cancer treatment education; Decision Tools
  Arms: the Information + Decision Aid group

SUMMARY:
We plan to test the effectiveness of a recently developed computer-based program that is designed to improve patient knowledge about prostate cancer treatments. It is also designed to help men clarify their values using a computer-based 'decision aid.' A decision aid gives patients tools to help them understand their own values and how these values may be related to their choice of different forms of therapy for prostate cancer. In order to test the effectiveness of the decision aid, men will be assigned on a chance basis to receive either 1) the computer program that includes the information about prostate cancer treatments alone, or 2) the computer program that contains both the information and the decision aid. We expect that men in decision aid group will be more active in their treatment decision and will have improved knowledge, quality of life, and satisfaction with the treatment decision relative to men who only receive the information.

DETAILED DESCRIPTION:
Background: There is a controversy in the medical community surrounding the utility of treatment options for clinically localized prostate cancer. Although several options are available for management of localized prostate cancer, no option is clearly superior to others. The main therapeutic options for localized prostate cancer include radical prostatectomy (RP), radiation therapy (RT; external beam radiation or brachytherapy), and expectant management (EM) or "watchful waiting." The American Urological Association, after a structured review of the available literature, concluded that there is insufficient evidence to clearly recommend RP, RT, or EM. They recommended that factors such as life expectancy, current health, and patient preference for therapeutic options be considered in the treatment decision. Since the survival benefits of the different management strategies are as of yet uncertain, and men's preferences for outcomes of therapy may influence the decision regarding management choice, men should be informed of potential outcomes and should be encouraged to examine their own values in deciding upon a management strategy for their prostate cancer.

Objective: The primary goal is to evaluate a method of patient education that is designed to provide treatment-related information and to help men clarify their preferences and values via a recently developed computer-based decision aid. We expect that men randomized to the decision aid condition will be more active in their treatment decision and will have improved patient outcomes relative to men assigned to the Information only condition.

Specific Aims. The specific aims are: 1) To evaluate the relative impact of providing newly diagnosed patients with computer-based prostate cancer treatment information vs. providing patients with the information plus an interactive decision-aid on a) shared decision-making practices and b) patient outcomes (decisional satisfaction, quality of life, knowledge), 2) To explore the mechanisms by which the decision aid impacts on SDM and patient outcomes, and 3) To identify men who are most and least likely to benefit from the education plus decision-aid intervention.

Study Design: Men will be accrued at the time of their biopsy and those with a positive biopsy result will receive the intervention following notification of the diagnosis but prior to their initial meeting with the urologist in which treatment options are discussed. Participants will be followed at one, six and twelve months post-intervention. The primary outcomes include patient outcomes (knowledge, quality of life, and decisional satisfaction) and shared decision making (SDM) practices.

Relevance In many areas of medicine, including treatment of localized prostate cancer, there has been a rapid expansion of research that has resulted in a growing number of diagnostic and treatment options that are available to physicians and patients. In many cases, there are several effective and viable treatment options, but randomized clinical trials assessing treatment effectiveness have not yet been completed. Although the availability of different options will undoubtedly be beneficial in the long run, at present it creates a difficult decision for individuals and physicians who are faced with the choices for which no best answer is known. The proposed study is designed to assist patient through this decision, by providing information and helping them to consider their values.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility criteria include: 1) ability to speak English, 2) absence of cognitive impairment that would limit participation in the study. 3) Diagnosis of localized prostate cancer. Participants will not be limited by age.

Exclusion Criteria:

* Men who have already made a treatment decision.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2002-09; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
treatment satisfaction, quality of life, prostate cancer knowledge at 1, 6, and 12 months post random assignment | one, six, and one year follow-up assesments

SECONDARY OUTCOMES:
shared decision making at 1, 6, and 12 months post random assignment. | one, six and one year follow-up assesments

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn L. Taylor, Ph.D., Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States